CLINICAL TRIAL: NCT01368588
Title: Androgen Deprivation Therapy and High Dose Radiotherapy With or Without Whole-Pelvic Radiotherapy in Unfavorable Intermediate or Favorable High Risk Prostate Cancer: A Phase III Randomized Trial
Brief Title: Androgen-Deprivation Therapy and Radiation Therapy in Treating Patients With Prostate Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-0924; CDR0000701128; NCI-2011-02674 (Registry Identifier: Clinical Trials Reporting Program (CTRP)); NCT02673190 (obsolete NCT alias)
Record Dates: First submitted 2011-06-07; First posted 2011-06-08 (Estimated); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage I prostate cancer; stage IIA prostate cancer; stage IIB prostate cancer; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Active Comparator): Patients undergo high-dose radiotherapy of the prostate and seminal vesicles using intensity-modulated radiotherapy (IMRT)* or 3D-conformal radiation therapy (3D-CRT)* once daily, 5 days a week, for approximately 9 weeks. Patients may also undergo permanent prostate implant (PPI) brachytherapy or high-dose rate brachytherapy (I 125 or Pd 103 may be used as the radioisotope).
  Interventions: Radiation: radiation therapy
- Arm II (Experimental): Patients undergo whole-pelvic radiotherapy (WPRT)* (3D-CRT or IMRT) once daily, 5 days a week, for approximately 9 weeks. Patients may also undergo brachytherapy as in arm I.
  Interventions: Radiation: Whole-pelvic radiotherapy (WPRT)

INTERVENTIONS:
Radiation: radiation therapy — Undergo RT using IMRT or 3D-CRT
  Arms: Arm I
Radiation: Whole-pelvic radiotherapy (WPRT) — Undergo whole-pelvic radiotherapy (WPRT)
  Arms: Arm II

SUMMARY:
RATIONALE: Androgens can cause the growth of prostate cancer cells. Androgen deprivation therapy may stop the adrenal glands from making androgens. Radiation therapy uses high-energy x-rays to kill tumor cells.

PURPOSE: This randomized phase III trial studies androgen-deprivation therapy and radiation therapy in treating patients with prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Demonstrate that prophylactic, neoadjuvant, androgen-deprivation therapy (NADT) and whole-pelvic radiation therapy (WPRT) will result in improvement in overall survival (OS) of patients with "unfavorable" intermediate-risk or "favorable" high-risk prostate cancer compared to NADT and high-dose prostate (P) and seminal vesicle (SV) radiation therapy (RT) using intensity-modulated RT (IMRT) or external-beam RT (EBRT) with a high-dose rate (HDR) or a permanent prostate (radioactive seed) implant (PPI) boost.

Secondary

* Demonstrate that prophylactic WPRT improves biochemical control.
* Determine the distant metastasis (DM)-free survival.
* Determine the cause-specific survival (CSS).
* Compare acute and late treatment-adverse events between patients receiving NADT and WPRT versus NADT, P, and SV RT.
* Determine whether health-related quality of life (HRQOL), as measured by the Expanded Prostate Cancer Index Composite (EPIC), significantly worsens with increasing aggressiveness of treatment (i.e., Arm 2, NADT + WPRT).
* Determine whether more aggressive treatment (Arm 2, NADT + WPRT) is associated with a greater increase in fatigue (PROMIS Fatigue Short Form) from baseline to last week of treatment, and a greater increase in circulating inflammatory markers (IL-1, IL-1ra, IL-6, tumor necrosis factor (TNF)-alpha, and C-reactive protein).
* Demonstrate an incremental gain in OS and CSS with more aggressive therapy that outweighs any detriments in the primary generic domains of HRQOL (i.e., mobility, self-care, usual activities, pain/discomfort, and anxiety/depression).
* Determine whether changes in fatigue from baseline to the next three time points (week prior to RT, last week of treatment, and 3 months after treatment) are associated with changes in circulating cytokines, mood, sleep, and daily activities across the same time points.
* Collect paraffin-embedded tissue blocks, plasma, whole blood, and urine for planned and future translational research analyses.

OUTLINE: This is a multicenter study. Patients are stratified according to moderate- to high-risk groups as listed in the Disease Characteristics of this abstract, type of radiotherapy boost (IMRT vs brachytherapy [Low-dose rate (LDR) using PPI or HDR]), and duration of androgen-deprivation therapy (short-term [6 months] vs long-term [32 months]). Patients are randomized to 1 of 2 treatment arms.

All patients receive neoadjuvant androgen-deprivation therapy comprising bicalutamide orally (PO) once daily or flutamide PO thrice daily for 6 months, and luteinizing hormone-releasing hormone (LHRH) agonist/antagonist therapy comprising leuprolide acetate, goserelin acetate, buserelin, triptorelin, or degarelix subcutaneously (SC) or intramuscularly (IM) every 1 to 3 months beginning 2 months prior to radiotherapy and continuing for 6 or 32 months.

Radiotherapy begins within 8 weeks after beginning LHRH agonist/antagonist injection.

* Arm I: Patients undergo high-dose radiotherapy of the prostate and seminal vesicles using intensity-modulated radiotherapy (IMRT)* or 3D-conformal radiation therapy (3D-CRT)* once daily, 5 days a week, for approximately 9 weeks. Patients may also undergo permanent prostate implant (PPI) brachytherapy or high-dose rate brachytherapy (iodine I 125 or palladium Pd 103 may be used as the radioisotope).
* Arm II: Patients undergo whole-pelvic radiotherapy (WPRT)* (3D-CRT or IMRT) once daily, 5 days a week, for approximately 9 weeks. Patients may also undergo brachytherapy as in arm I.

NOTE: * Patients undergoing brachytherapy implant receive 5 weeks of IMRT, 3D-CRT, or WPRT.

Patients may undergo blood and urine sample collection for correlative studies. Primary tumor tissue samples may also be collected.

Patients may complete the Expanded Prostate Cancer Index Composite (EPIC), the PROMIS-Fatigue Short Form, and the EuroQol (EQ-5D) quality-of-life (QOL) questionnaires at baseline and periodically during treatment. Patients who participate in the QOL portion of the study must also agree to periodic blood collection.

After completion of study therapy, patients are followed up every 3 months for 1 year, every 6 months for 3 years, and then yearly thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Pathologically (histologically or cytologically) proven diagnosis of prostatic adenocarcinoma within 180 days of registration at moderate- to high-risk for recurrence as determined by one of the following combinations:

  * Gleason score 7-10 + T1c-T2b (palpation) + prostate-specific antigen (PSA) < 50 ng/mL (includes intermediate- and high-risk patients)
  * Gleason score 6 + T2c-T4 (palpation) + PSA < 50 ng/mL OR
  * Gleason score 6 + >= 50% (positive) biopsies + PSA < 50 ng/ml
  * Gleason score 6 + T1c-T2b (palpation) + PSA > 20 ng/mL Patients previously diagnosed with low risk prostate cancer undergoing active surveillance who are re-biopsied and found to have unfavorable intermediate risk disease or favorable high risk disease according to the protocol criteria are eligible for enrollment within 180 days of the repeat biopsy procedure.
* History and/or physical examination (to include at a minimum digital rectal examination of the prostate and examination of the skeletal system and abdomen) within 90 days prior to registration
* Clinically negative lymph nodes as established by imaging (pelvic and/or abdominal CT or MR), (but not by nodal sampling, or dissection) within 90 days prior to registration

  * Patients with lymph nodes equivocal or questionable by imaging are eligible if the nodes are ≤ 1.5 cm
  * Patients status post a negative lymph node dissection are not eligible
* No evidence of bone metastases (M0) on bone scan within 120 days prior to registration (Na F PET/CT is an acceptable substitute)

  * Equivocal bone scan findings are allowed if plain films (or CT or MRI) are negative for metastasis
* Baseline serum PSA value performed with an FDA-approved assay (e.g., Abbott, Hybritech) within 120 days prior to registration
* Study entry PSA should not be obtained during the following time frames:

  * Ten-day period following prostate biopsy
  * Following initiation of hormonal therapy
  * Within 30 days after discontinuation of finasteride
  * Within 90 days after discontinuation of dutasteride

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-1
* Absolute neutrophil count (ANC) ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin (Hgb) ≥ 8.0 g/dL (transfusion or other intervention to achieve Hgb ≥ 8.0 g/dL is acceptable)
* No prior invasive (except non-melanoma skin cancer) malignancy unless disease-free for a minimum of 3 years (1,095 days) and not in the pelvis

  * E.g., carcinoma in situ of the oral cavity is permissible; however, patients with prior history of bladder cancer are not allowed
  * No prior hematological (e.g., leukemia, lymphoma, or myeloma) malignancy
  * No previous radical surgery (prostatectomy) or cryosurgery for prostate cancer
  * No previous pelvic irradiation, prostate brachytherapy or bilateral orchiectomy
  * No previous hormonal therapy, such as LHRH agonists (e.g., leuprolide, goserelin, buserelin, triptorelin) or LHRH antagonist (e.g. degarelix), anti-androgens (e.g., flutamide, bicalutamide, cyproterone acetate), estrogens (e.g., DES), or surgical castration (orchiectomy)
* Prior pharmacologic androgen ablation for prostate cancer is allowed only if the onset of androgen ablation (both LHRH agonist and oral anti-androgen) is ≤ 45 days prior to the date of registration.
* No severe, active co-morbidity, defined as any of the following:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
  * Transmural myocardial infarction within the last 6 months
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects or severe liver dysfunction
  * Acquired immune deficiency syndrome (AIDS) based upon current Centers for Disease Control (CDC) definition

    * Protocol-specific requirements may also exclude immuno-compromised patients
    * HIV testing is not required for entry into this protocol
* No patients who are sexually active and not willing/able to use medically acceptable forms of contraception
* No prior allergic reaction to the hormones involved in this protocol

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior radical surgery (prostatectomy) or cryosurgery for prostate cancer
* No prior pelvic irradiation, prostate brachytherapy, or bilateral orchiectomy
* No prior hormonal therapy, such as luteinizing hormone-releasing hormone (LHRH) agonists (e.g., leuprolide, goserelin, buserelin, triptorelin) or LHRH antagonist (e.g., degarelix), anti-androgens (e.g., flutamide, bicalutamide, cyproterone acetate), estrogens (e.g., diethylstilbestrol (DES) ), or surgical castration (orchiectomy)
* No prior pharmacologic androgen ablation for prostate cancer unless the onset of androgen ablation is ≤ 45 days prior to the date of registration
* No finasteride within 30 days prior to registration
* No dutasteride or dutasteride/tamsulosin (Jalyn) within 90 days prior to registration
* No prior or concurrent cytotoxic chemotherapy for prostate cancer

  * Prior chemotherapy for a different cancer is allowable
* No prior radiotherapy, including brachytherapy, to the region of the study cancer that would result in overlap of radiation therapy fields

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2592 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2025-04-17 (Actual); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | From date of randomization to the date of death.

SECONDARY OUTCOMES:
Cause-specific survival | From date of randomization to the date of death due to prostate cancer.
Distant metastasis-free survival | From date of randomization to the date of first documented distant metastasis or date of first clinical and/or radiographic appearance of disseminated disease.
Biochemical failure by the Phoenix definition (PSA ≥ 2 ng/mL over the nadir PSA) | From date of randomization to the date of first biochemical failure by phoenix definition within 5 years of randomization.
Incidence of "acute" adverse events as assessed by the Common Toxicity Criteria for Adverse Effects (CTCAE) current version | From protocol treatment start date to the date of first occurrence of worst severity of the adverse event </= 30 days from completion of radiation therapy.
Time to "late" grade 3+ adverse events as assessed by CTCAE current version | From protocol treatment start date to the date of the first late grade 3+ adverse event occurring more than 30 days after the completion of radiation therapy.
Prostate cancer-specific HRQOL change as measured by the EPIC-26 (bowel or urinary domain) | Date when baseline EPIC-26 completed to 6 months post radiation therapy, 1 year post radiation therapy and 5 years post radiation therapy.
Fatigue status as measured by the Patient-Reported Outcome Measurement Information System (PROMIS) fatigue-domain change score | From the date when the baseline PROMIS is completed to the last week of treatment.
Assessment and comparison of Quality Adjusted Life Years (QALYs) | From the baseline QALYs assessment to the last week of radiation therapy (RT), 3 months post RT, 6 months post RT, 1 year post RT and 5 years post RT.

CONTACTS AND LOCATIONS:
Overall Officials: Mack Roach, MD, Principal Investigator — University of California, San Francisco
Locations (478):
- United States (454):
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Arizona Breast Cancer Specialists-Gilbert, Gilbert, Arizona
  - Arizona Center for Cancer Care-Peoria, Peoria, Arizona
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Saint Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Arizona Breast Cancer Specialists-Phoenix, Phoenix, Arizona
  - Arizona Oncology-Deer Valley Center, Phoenix, Arizona
  - 21st Century Oncology-Scottsdale, Scottsdale, Arizona
  - Arizona Breast Cancer Specialists, Scottsdale, Arizona
  - Arizona Breast Cancer Specialists-Scottsdale, Scottsdale, Arizona
  - Arizona Oncology Services Foundation, Scottsdale, Arizona
  - Arizona Center for Cancer Care-Surprise, Surprise, Arizona
  - Arizona Oncology Associates-West Orange Grove, Tucson, Arizona
  - University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - AIS Cancer Center at San Joaquin Community Hospital, Bakersfield, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Mercy San Juan Medical Center, Carmichael, California
  - Adventist Health Cancer Care Center Chico, Chico, California
  - Fresno Cancer Center, Fresno, California
  - Saint Agnes Medical Center, Fresno, California
  - Marin General Hospital, Greenbrae, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Tibor Rubin VA Medical Center, Long Beach, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Mercy UC Davis Cancer Center, Merced, California
  - Memorial Medical Center, Modesto, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Desert Regional Medical Center, Palm Springs, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Pomona Valley Hospital Medical Center, Pomona, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Santa Clara Valley Medical Center, San Jose, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Saint Joseph's Medical Center, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Shaw Cancer Center, Edwards, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Hartford HealthCare - Saint Vincent's Medical Center, Bridgeport, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Middlesex Hospital, Middletown, Connecticut
  - Helen F Graham Cancer Center, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Broward Health North, Deerfield Beach, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Baptist Medical Center South, Jacksonville, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Cancer Center of Putnam, Palatka, Florida
  - GenesisCare USA - Plantation, Plantation, Florida
  - James A. Haley Veterans Affairs Hospital, Tampa, Florida
  - Florida Cancer Affiliates, Trinity, Florida
  - Cleveland Clinic-Weston, Weston, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Central Georgia Gynecologic Oncology, Macon, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Queen's Medical Center, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Rush - Copley Medical Center, Aurora, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Weiss Memorial Hospital, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - UChicago Medicine Comprehensive Cancer Center - Saint Joseph Hospital, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - SwedishAmerican Regional Cancer Center/ACT, Rockford, Illinois
  - Saint John's Hospital, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Radiation Oncology Associates PC, Fort Wayne, Indiana
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - McFarland Clinic PC - Ames, Ames, Iowa
  - Saint Luke's Hospital, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Finley Hospital, Dubuque, Iowa
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Saint Catherine Hospital, Garden City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Olathe Health Cancer Center, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Owensboro Health Mitchell Memorial Cancer Center, Owensboro, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Covington, Covington, Louisiana
  - Mary Bird Perkins Cancer Center - Houma, Houma, Louisiana
  - East Jefferson General Hospital, Metairie, Louisiana
  - LSU Healthcare Network / Metairie Multi-Specialty Clinic, Metairie, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Touro Infirmary, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Anne Arundel Medical Center, Annapolis, Maryland
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Saint Agnes Hospital, Baltimore, Maryland
  - UM Upper Chesapeake Medical Center, Bel Air, Maryland
  - Central Maryland Radiation Oncology in Howard County, Columbia, Maryland
  - University of Maryland Radiation Oncology Center at Union Hospital, Elkton, Maryland
  - UM Baltimore Washington Medical Center/Tate Cancer Center, Glen Burnie, Maryland
  - TidalHealth Peninsula Regional, Salisbury, Maryland
  - UM Saint Joseph Medical Center, Towson, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Saint Anne's Hospital, Fall River, Massachusetts
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Beth Israel Deaconess Hospital-Plymouth, Plymouth, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Veteran's Administration Medical Center - Ann Arbor, Ann Arbor, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - McLaren Cancer Institute-Bay City, Bay City, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - GenesisCare USA - Clarkston, Clarkston, Michigan
  - McLaren Cancer Institute-Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Beaumont Hospital - Dearborn, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - GenesisCare USA - Farmington Hills, Farmington Hills, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Beaumont Hospital - Farmington Hills, Farmington Hills, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Karmanos Cancer Institute at McLaren Greater Lansing, Lansing, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - McLaren Cancer Institute-Lapeer Region, Lapeer, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - McLaren Cancer Institute-Central Michigan, Mount Pleasant, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - McLaren Cancer Institute-Owosso, Owosso, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - 21st Century Oncology-Pontiac, Pontiac, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - McLaren-Port Huron, Port Huron, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - GenesisCare USA - Troy, Troy, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Mayo Clinic Health System in Albert Lea, Albert Lea, Minnesota
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Mayo Clinic Health Systems-Mankato, Mankato, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Freeman Health System, Joplin, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Kansas City Veterans Affairs Medical Center, Kansas City, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Veteran's Affairs Medical Center - Saint Louis, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Renown Regional Medical Center, Reno, Nevada
  - Exeter Hospital, Exeter, New Hampshire
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - AtlantiCare Surgery Center, Egg Harbor, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Inspira Medical Center Mullica Hill, Mullica Hill, New Jersey
  - Penn Medicine Princeton Health, Plainsboro, New Jersey
  - Sidney Kimmel Cancer Center Washington Township, Sewell, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Sparta Cancer Treatment Center, Sparta, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - Memorial Medical Center - Las Cruces, Las Cruces, New Mexico
  - South Shore University Hospital, Bay Shore, New York
  - New York-Presbyterian/Brooklyn Methodist Hospital, Brooklyn, New York
  - Sands Cancer Center, Canandaigua, New York
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Arnot Ogden Medical Center/Falck Cancer Center, Elmira, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Wilmot Cancer Institute Radiation Oncology at Greece, Rochester, New York
  - Highland Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - James J Peters VA Medical Center, The Bronx, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Durham VA Medical Center, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - The Coleman Radiation Center-Carteret General Hospital, Morehead City, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - UNC Rex Cancer Center, Raleigh, North Carolina
  - NHRMC Radiation Oncology - Supply, Supply, North Carolina
  - NHRMC Radiation Oncology - 16th Street, Wilmington, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - Cleveland Clinic Akron General, Akron, Ohio
  - Summa Health System - Barberton Campus, Barberton, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Cleveland Clinic Mercy Hospital, Canton, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Summa Health Medina Medical Center, Medina, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - University Hospitals Portage Medical Center, Ravenna, Ohio
  - UH Seidman Cancer Center at Salem Regional Medical Center, Salem, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - University of Toledo, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Saint John Medical Center, Tulsa, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Three Rivers Community Hospital, Grants Pass, Oregon
  - Providence Medford Medical Center, Medford, Oregon
  - Rogue Valley Medical Center, Medford, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Northeast Radiation Oncology Center, Dunmore, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Fox Chase Cancer Center Buckingham, Furlong, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Cherry Tree Cancer Center, Hanover, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - Upper Delaware Valley Cancer Center, Milford, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Tidelands Georgetown Memorial Hospital, Georgetown, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - The Radiation Oncology Center-Hilton Head/Bluffton, Hilton Head Island, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Erlanger Medical Center, Chattanooga, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Texas Cancer Center, Abilene, Texas
  - Texas Oncology PA Beaumont, Beaumont, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Texas Oncology - Denison Cancer Center, Denison, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Texas Oncology - Fort Worth Cancer Center, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Memorial Hermann Memorial City Medical Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - UTMB Cancer Center at Victory Lakes, League City, Texas
  - Texas Oncology-McAllen, McAllen, Texas
  - Texas Oncology-McKinney, McKinney, Texas
  - West Texas Cancer Center, Odessa, Texas
  - Texas Oncology-Plano West, Plano, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Texas Oncology Cancer Center Sugar Land, Sugar Land, Texas
  - Deke Slayton Cancer Center, Webster, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Ogden Regional Medical Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - Southwestern Vermont Medical Center, Bennington, Vermont
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - Norris Cotton Cancer Center-North, Saint Johnsbury, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Augusta Health Center for Cancer and Blood Disorders, Fishersville, Virginia
  - Sentara Cancer Institute at Sentara CarePlex Hospital, Hampton, Virginia
  - Sentara Rockingham Memorial Hospital Hahn Cancer Center, Harrisonburg, Virginia
  - Bon Secours DePaul Medical Center, Norfolk, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Hunter Holmes McGuire Veterans Administration Medical Center, Richmond, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Roanoke, Virginia
  - Sentara Obici Hospital, Suffolk, Virginia
  - Sentara Virginia Beach General Hospital, Virginia Beach, Virginia
  - Saint Francis Hospital, Federal Way, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - United Hospital Center, Bridgeport, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - ThedaCare Regional Medical Center - Appleton, Appleton, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Elmbrook Campus, Brookfield, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Mayo Clinic Health System Eau Claire Hospital-Luther Campus, Eau Claire, Wisconsin
  - Ascension Saint Francis - Reiman Cancer Center, Franklin, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - UW Cancer Center Johnson Creek, Johnson Creek, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Ascension Columbia Saint Mary's Hospital Ozaukee, Mequon, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Saint Joseph Campus, Milwaukee, Wisconsin
  - Ascension Columbia Saint Mary's Hospital - Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Zablocki Veterans Administration Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Ascension All Saints Hospital, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Clinic Stevens Point Center, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
  - Billings Clinic-Cody, Cody, Wyoming
- Canada (18):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA-Cancer Centre for the Southern Interior, Kelowna, British Columbia
  - BCCA-Fraser Valley Cancer Centre, Surrey, British Columbia
  - Doctor H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - QEII Health Sciences Centre/Nova Scotia Health Authority, Halifax, Nova Scotia
  - London Regional Cancer Program, London, Ontario
  - Stronach Regional Health Centre at Southlake, Newmarket, Ontario
  - Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - McGill University Department of Oncology, Montreal, Quebec
  - CHUM - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - The Research Institute of the McGill University Health Centre (MUHC), Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - CHU de Quebec-L'Hotel-Dieu de Quebec (HDQ), Québec, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Pamela Youde Nethersole Eastern Hospital, Chai Wan, Hong Kong
- Israel (2):
  - Rabin Medical Center, Petah Tikva
  - Chaim Sheba Medical Center, Tel Litwinsky
- Singapore (2):
  - National University Hospital Singapore, Singapore
  - National Cancer Centre Singapore, Singapore
- Kantonsspital Aarau, Aarau, Switzerland

IPD SHARING:
Plan to Share IPD: No